CLINICAL TRIAL: NCT06311227
Title: A Phase 2 Study of Venetoclax in Relapsed Classic or Variant Hairy Cell Leukemia
Brief Title: Venetoclax for the Treatment of Patients With Relapsed Hairy Cell Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01904; NCI-2024-01904 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10637 (Other: National Cancer Institute LAO); 10637 (Other: CTEP)
Record Dates: First submitted 2024-03-13; First posted 2024-03-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Hairy Cell Leukemia; Recurrent Hairy Cell Leukemia Variant
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Specimen Handling; Biopsy; Spinal Puncture; Magnetic Resonance Spectroscopy; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI and blood sample collection throughout the study. Patients may undergo bone marrow biopsy and/or aspiration on study. Additionally, patients with known or suspected CNS disease undergo lumbar puncture throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests how well venetoclax works in treating patients with hairy cell leukemia that has come back after a period of improvement (relapsed). Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR) of venetoclax.

SECONDARY OBJECTIVES:

I. To determine the complete remission (CR) and minimal residual disease (MRD)-negative CR rates of venetoclax in relapsed hairy cell leukemia/hairy cell leukemia variant (HCL/HCLv).

II. To determine the rates of MRD-negative by blood flow cytometry with venetoclax.

III. To determine the safety of venetoclax in relapsed HCL/HCLv. IV. To determine the response and CR duration and MRD-negative survival in relapsed HCL/HCLv receiving venetoclax.

EXPLORATORY OBJECTIVES:

I. To correlate response to TP53 mutations and other mutations, particularly for BRAF wild-type (WT) relapsed HCL/HCLv.

II. To perform whole exome sequencing (WES) of relapsed HCL/HCLv samples to look for mutations, to correlate with response.

OUTLINE:

Patients receive venetoclax orally (PO) once daily (QD) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the study. Patients may undergo bone marrow biopsy and/or aspiration on study. Additionally, patients with known or suspected central nervous system (CNS) disease undergo lumbar puncture throughout the study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed HCL/HCLv after purine analog therapy who are relapsed from or are ineligible for BRAF therapy and have not received prior venetoclax
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Total bilirubin ≤ 3 x institutional upper limit of normal (ULN) unless consistent with Gilbert's (ration between total and direct bilirubin > 5)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN
* Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 45 mL/min/1.73m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have had no HCL/HCLv treatment for ≥ 4 weeks prior to enrollment, and those with treatment > 4 weeks prior to enrollment must not be responding to their last treatment with decreasing tumor burden or improving disease related cytopenias
* Patients must have a need for treatment due to absolute neutrophil count (ANC) < 1/nL, hemoglobin (Hgb) < 10g/dL, platelets (Plt) < 100/nL, symptomatic splenomegaly, HCL mass with short axis > 2cm outside or > 0.5 cm inside the CNS, HCL/HCLv count > 5/nL in blood or > 25/mm^3 in cerebrospinal fluid (CSF), HCL/HCLv doubling time < 6 months and increasing lytic or blastic bone lesions
* The effects of venetoclax on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during treatment and for 30 days after the last dose of venetoclax. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception during treatment and for 30 days after the last dose of venetoclax
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Ability and willingness to swallow pills

Exclusion Criteria:

* Patients who have received prior venetoclax
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to venetoclax
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because venetoclax is a B-cell lymphoma-2 (BCL-2) inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, breastfeeding should be discontinued if the mother is treated with venetoclax
* Malabsorption syndrome or other conditions that would interfere with intestinal absorption
* Live attenuated vaccines should not be administered within 4 weeks prior to, during, or 30 days after study treatment and recovery has occurred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 30 days after the last dose
  Will be determined with 95% confidence intervals for each group.

SECONDARY OUTCOMES:
Complete remission (CR) rate | Up to 30 days after the last dose
  CR will be defined as resolution of cytopenias with neutrophils > 1.5/nL, platelets > 100/nL, and hemoglobin > 11g/dL at least 4 weeks from last transfusion or growth factor, resolution of splenomegaly by exam or by spleen size =< 17 cm by imaging, resolution of hairy cell leukemia (HCL)/hairy cell leukemia variant (HCLv)-related lymphadenopathy/masses to =< 2cm in short axis (=< 0.5 cm in short axis in the central nervous system [CNS]), and absence of morphological evidence of HCL/HCLv in the blood and bone marrow.
Minimal residual disease (MRD)-negative CR rate | Up to 30 days after the last dose
  Defined as meeting the criteria for CR plus absence of HCL/HCLv cells in the bone marrow aspirate and blood by flow cytometry, and negative immunochemistry of the bone marrow biopsy. Positive IHC involves B-cells > T-cells and most of the B-cells being consistent with HCL. Patients with CNS disease who achieve CR with positive cerebrospinal fluid flow cytometry will be considered CR with MRD.
MRD negativity | Up to 30 days after the last dose
  Will determine the rates of MRD-negative by blood flow cytometry.
Incidence of adverse events | Up to 30 days after the last dose
Complete response duration | Up to 30 days after the last dose
MRD-negative survival | Up to 30 days after the last dose

OTHER OUTCOMES:
TP53 mutations and other mutations | Up to 30 days after the last dose
  Will correlate response to TP53 mutations and other mutations.
Whole exome sequencing of relapsed HCL/HCLv samples | Up to 30 days after the last dose
  Will perform whole exome sequencing of relapsed HCL/HCLv samples to look for mutations, to correlate with response.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, Principal Investigator — National Cancer Institute LAO
Locations (21):
- United States (21):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm